CLINICAL TRIAL: NCT07134387
Title: BronQ Family: Assessing the Long-term Impact of Bronchopulmonary Dysplasia (BPD) on Affected Families' Health-related Quality of Life
Brief Title: Long-Term Burden of BPD and Health-Related Quality of Life (BronQ Family)
Acronym: BronQ Family
Status: Recruiting | Type: Observational
Sponsor: Global Foundation for the Care of Newborn Infants (Other)
Collaborators: European Society for Paediatric Research (ESPR) (Unknown); Union of European Neonatal and Perinatal Societies (UENPS) (Unknown); European Respiratory Society (ERS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: METC 2025-0285
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Bronchopulmonary Dysplasia (BPD); Chronic Lung Disease of Newborn; HRQOL (Health Related Quality Of Life)
Keywords: Parental Quality of life; QoL; Health-related quality of life; HRQoL; Caregiver burden; Parental well-being; Family; Bronchopulmonary Dysplasia (BPD); Chronic Lung Disease (CLD); Chronic Lung Diseaseof Newborn; Respiratory Morbidity; Long-term outcomes; Parents; Caregivers; Infants; Newborn; Children; Preterm; Prematurity; NICU; Intensive Care; Neonatal; Survey; Questionnaire; Multinational study; retrospective data collection; participatory research; Patient-reported outcomes; PROs; Patient-reported outcome measures; PROMs
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Caregiver Burden; Premature Birth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents or caregivers of children with (a history of) physician diagnosed BPD: The primary population of this study consists of parents and caregivers of preterm born children (< 37 weeks of gestation) under 18 years old who have been diagnosed with newborn-onset Bronchopulmonary Dysplasia (BPD). Furthermore, the child should have been discharged from their initial hospital stay after birth. Participants will be recruited from multiple countries, including France, Germany, Italy, the Netherlands, Spain, the United Kingdom (including Northern Ireland), and the United States.
  Interventions: Other: N/A, no intervention, participation in survey
- Parents or caregivers of preterm born children without chronic health conditions: The control group consists of parents and caregivers of preterm born children (< 37 weeks of gestation) under 18 years old who do not report a history of BPD. Furthermore, the child should have been discharged from their initial hospital stay after birth. They will as well be recruited from France, Germany, Italy, the Netherlands, Spain, the United Kingdom (including Northern Ireland), and the United States. If the final sample size permits, a post hoc filter will be applied to restrict analyses to the subgroup of very preterm (< 32 weeks gestation) and/or very low birthweight (< 1500 g birthweight) children.
  Interventions: Other: N/A, no intervention, participation in survey

INTERVENTIONS:
Other: N/A, no intervention, participation in survey — A unified questionnaire will be utilized for all participants, irrespective of their group assignment. Participants will be assigned to the BPD or comparison group retrospectively, based on their answers defining the BPD-status. To enhance comprehension, the questionnaire avoids using the term "BPD" wherever feasible and instead employs a more general reference to lung problems.

SUMMARY:
The objective of this study is to examine the long-term impact of having a child with Bronchopulmonary Dysplasia (BPD) on the parents and caregivers from the time of diagnosis through adulthood. The primary focus will be on parents and caregivers of children until the age of 18 (< 18) years who were diagnosed with BPD as newborns. Data will be collected through an online questionnaire in France, Germany, Italy, the Netherlands, Spain, the United Kingdom (including Northern Ireland), and the United States. It will ask about inclusion and exclusion criteria, background information (caregiver, child, and family situation), the child's medical situation, parental health-related quality of life (HRQoL), health literacy, feelings, support structures, and economic burden of the family.

DETAILED DESCRIPTION:
The study will be designed as an observational, cross-sectional survey with a comparison group using a self-administered, web-based questionnaire for retrospective data collection. The study will use a multi-lingual online survey collecting data from parents in France, Germany, Italy, the Netherlands, Spain, the United Kingdom (including Northern Ireland), and the United States. Following a participatory research approach, the study will be carried out in close collaboration with representatives of national and international parent organizations, affected parents and/or former patients, professional healthcare societies, healthcare professionals as well as health researchers in the form of a Project Expert Group (PEG). It includes medical experts in BPD and neonatal/pediatric care, parent representatives, and, if applicable, parents of children affected by BPD during the neonatal period and/or affected patients from the countries of interest. The PEG will be complemented by the External Scientific Advisory Board (ESAB), which comprises n=4 members, including researchers specializing in HRQoL and/or pediatric respiratory outcomes research, including BPD. The PEG and ESAB will be engaged in all stages of the research project through regular online meetings. The ESAB contributes mainly to the study design and conception, questionnaire development, data analysis and interpretation, and will support the development of scientific publications. The remaining members of the PEG are involved in reviewing all final materials generated from the project and support the recruitment of study participants, as well as the dissemination of findings within their professional networks.

After comprehensive literature research and exchange with the study experts, the questionnaire will be drafted considering the already existing PedsQL Family Impact Module (FIM) (15) to assess parental HRQoL. In addition to socio-demographic information and inclusion/exclusion criteria, the questionnaire includes items evaluating various dimensions of parental HRQoL, health literacy and support structures. Furthermore, questions assessing the child's medical situation, treatment and eventual co-morbidities during the newborn period as well as at the time of the current survey will be added. Ultimately, questions addressing the financial burden of medical costs will be considered to assess the personal impact as well as the impact on the healthcare system in the respective countries. A unified questionnaire will be utilized for all participants, irrespective of their group assignment. Participants will be assigned to the BPD or comparison group retrospectively, based on their answers defining the BPD-status. To enhance comprehension, the questionnaire avoids using the term "BPD" wherever feasible and instead employs a more general reference to lung problems.

The questionnaire draft will be developed in close collaboration with the ESAB and reviewed by the PEG. After implementing necessary changes, the updated version will be shared again with the expert groups for final review. In addition, a pretest with up to 10 participants resembling the target group will be performed to elaborate on understanding, relevance and completeness as well as to elucidate other relevant topics that have not yet been covered and still need to be included.

After a potential adaptation based on data and information of the pre-testing, the questionnaire will be translated in the respective country languages with the PEG reviewing the translations. The translated questionnaire versions will be transferred into the online survey software SurveyMonkey® and will be distributed via the PEG/ESAB, GFCNI's network, GFCNI's newsletter and social media channels via an access link.

GFCNI received a research grant from Chiesi in support of this independent study.

ELIGIBILITY:
Inclusion Criteria:

BPD-group:

* Being a parent or primary caregiver of a child until the age of 18 years (0 to under 18 years),

  * who was born preterm (before 37 weeks of gestation),
  * who has been discharged from their initial hospital stay after birth,
  * who suffered from BPD in the newborn period and
  * who was born or is currently living in the following countries: France, Germany, Italy, the Netherlands, Spain, the United Kingdom (including Northern Ireland) and the United States
* providing sufficient proficiency in one of the languages of the questionnaire

Control group:

* Being a parent or primary caregiver of a child until the age of 18 years (0 to under 18 years),

  * who was born preterm (before 37 weeks of gestation),
  * who has been discharged from their initial hospital stay after birth,
  * who did not suffer from BPD in the newborn period and
  * who was born or is currently living in the following countries: France, Germany, Italy, the Netherlands, Spain, the United Kingdom (including Northern Ireland) and the United States
* providing sufficient proficiency in one of the languages of the questionnaire

Exclusion Criteria:

BPD-group:

* Other family members than parents/primary caregivers
* Parents or primary caregivers

  * of a child older/equal than 18 years of age
  * of a child with BPD who has not been discharged yet
  * of a child without a BPD in the newborn period
  * with insufficient proficiency in one of the languages available in the questionnaire

Control group:

* Other family members than parents/primary caregivers
* Parents or primary caregivers

  * of children older/equal than 18 years of age
  * of a child born term
  * of a child without BPD who has not been discharged yet
  * with insufficient proficiency in one of the languages available in the questionnaire

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consists of parents and caregivers of preterm-born children under 18 years old who have already been discharged from their initial hospital stay. Participants will be recruited from multiple countries, including France, Germany, Italy, the Netherlands, Spain, the United Kingdom/Northern Ireland, and the United States. They will be assigned to the BPD or comparison group retrospectively, based on their answers defining the BPD-status.
Sampling Method: Non-Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Parental health-related quality of life (HRQoL) assesed by Pediatric Quality of Life Inventory, Family Impact Module (PedsQL FIM) | 09/2025 - 02/2026
  To record the parents' HRQoL, the Pediatric Quality of Life Inventory Family Impact Module (PedsQL FIM) is implemented, a validated and widely used instrument designed to measure the impact of pediatric acute and chronic health conditions on parents and the family. It consists of 36 items across six parental dimensions (physical, emotional, social, and cognitive functioning, communication, and worry), as well as family daily activities and relationships. It is validated in all official languages of the seven participating countries (English, French, German, Italian, Dutch, Spanish) and allows the calculation of a sum score.

SECONDARY OUTCOMES:
Participant characteristics assesed by self developed online questionnaire | 09/2025 - 02/2026
  Inclusion/exclusion criteria, Baseline characteristics, socio-demographic characteristics of parent/caregiver, child, and the family situation
Medical Situation of the child assesed by self developed online questionnaire (parent report) | 09/2025 - 02/2026
  The section assesses the child's overall health, daily functioning, school attendance, and involvement of medical specialists. It covers emotional, cognitive, and behavioral issues (potentially linked to BPD), respiratory health (symptoms, infections, treatments, support), and feeding difficulties. It also records comorbidities and developmental impairments, and includes questions on RSV prevention and infection history.
Economic burden on families (Quantitative and qualitative) assesed by adapted version of the Family Economic Impact Inventory (Domain Family Finances) | 09/2025 - 02/2026
  The Family Finances section captures family costs related to caring for a child with health conditions, including direct and broader economic impacts such as financial burden, work productivity loss, and healthcare utilization.
Health Literacy (Quantitative) assesed by self-developed online questionnaire | 09/2025 - 02/2026
  Disease awareness and awareness of consequences
Support Structures (Quantitative and qualitative) assesed by self developed online questionnaire | 09/2025 - 02/2026

CONTACTS AND LOCATIONS:
Overall Officials: Julia Feiler, Dr, Principal Investigator — Global Foundation for the Care of Newborn Infants (GFCNI)
Locations (1):
- Global Foundation for the Care of Newborn Infants (GFCNI), München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No